CLINICAL TRIAL: NCT05312307
Title: Strata EXPress™: A Study Using StrataEXP™ to Identify RNA-Expression Biomarkers in Advanced Cancer Patients
Acronym: StrataEXPress
Status: Withdrawn | Type: Observational
Why Stopped: Screening of RNA expression profiles will be integrated directly into the Strata PATH study.
Sponsor: Strata Oncology (Industry)
Responsible Party: Sponsor
Other Study IDs: STR-006-001
Record Dates: First submitted 2022-03-26; First posted 2022-04-05 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary goal of this study is to identify patients with RNA expression profiles consistent with eligibility requirements for therapeutic clinical trials across solid tumors. Left-over tumor tissue will be collected from eligible participants for RNA expression analysis using next-generation sequencing.

DETAILED DESCRIPTION:
The primary goal of this study is to identify patients with RNA expression profiles consistent with eligibility requirements for therapeutic clinical trials across solid tumors. Left-over tumor tissue will be collected from eligible participants for RNA expression analysis using next-generation sequencing.

A parallel study, StrataPATH™ (STR-004-001), has been developed to support therapeutic hypotheses. Participants may be consented and screened for enrollment separately into StrataPATH with an eligible matching biomarker/drug treatment cohort upon positive identification of a relevant expression signature. Treatment effectiveness of antibody drug conjugates and other targeted therapies will be evaluated in these molecularly defined cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥18 years of age,
2. Participant must have pathologically confirmed advanced, metastatic, or recurrent solid tumor,
3. Measurable disease,
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2,
5. Participant must meet at least 1 of the following:

   1. Is/has not adequately responded to standard therapy, or
   2. For whom no life-extending standard therapy exists, or
   3. Who decline standard therapy, or
   4. In the opinion of the investigator, is not a candidate for or would be unlikely to tolerate or derive significant clinical benefit from standard therapy
6. Adequate cardiac, bone marrow, organ function & laboratory parameters as determined by the treating physician for potential participation in a clinical trial,
7. Leftover formalin-fixed, paraffin-embedded (FFPE) tumor tissue available for StrataEXP testing

Exclusion Criteria:

1. Females who are pregnant or nursing,
2. History of stroke including transient ischemic attack (TIA) or acute myocardial infarction within 4 months of enrollment,
3. Any other clinically significant medical condition that, in the opinion of the treating physician, makes participation in a clinical trial undesirable, including but not limited to ongoing or active infection, significant uncontrolled hypertension, or severe psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are male or female ≥ 18 years of age; must have pathologically confirmed advanced, metastatic, or recurrent solid tumor; measurable disease; have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2; must meet at least 1 of the following: a. Is/has not adequately responded to standard therapy, or b. For whom no life extending standard therapy exists, or c. Who decline standard therapy, or d. In the opinion of the investigator, is not a candidate for or would be unlikely to tolerate or derive significant clinical benefit from standard therapy; have adequate cardiac, bone marrow, organ function & laboratory parameters as determined by the treating physician for potential participation in a clinical trial; have leftover formalin-fixed, paraffin-embedded (FFPE) tumor tissue available for StrataEXP testing.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
To identify subjects with RNA signatures who may be eligible for clinical trial enrollment | 5 years
  The percentage of participants identified as eligible for therapeutic clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Kat Kwiatkowski, PhD, Study Director — Strata Oncology

IPD SHARING:
Plan to Share IPD: No